CLINICAL TRIAL: NCT07031310
Title: Correlation Between Forward Head Posture and Cervical Radiculopathy in Smart Phone Users
Brief Title: Correlation Between Forward Head Posture and Cervical Radiculopathy
Status: Enrolling by invitation | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Rafat, Assistant professor of physical therapy, Cairo University
Other Study IDs: P.T.REC/025/00087
Record Dates: First submitted 2025-06-11; First posted 2025-06-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-06

CONDITIONS: Smart Phone Users
Keywords: Forward head posture; Cervical Radiculopathy; Smart phone users
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- smart phone users

SUMMARY:
The progression rate of forward head posture has increased because of the increase in postural loads, to which individuals are subjected because of developed technologies including mobile phones, computers, and televisions. Postural abnormality in the upper cervical region has the potential to lead to nerve irritation and cervical radiculopathy. so the purpose of study is to investigate if there is a relationship between forward head posture and cervical radiculopathy in smart phone users.

DETAILED DESCRIPTION:
Cross-sectional observational study . 120 Participants will be recruited from students and employees of Nahda university (smart phone users) from both genders with age ranged between (18-35) years old.

outcomes measurement

1. Photogrammetric method to assess CVA by smart phone application FHP
2. Smartphone application for measuring cervical range of motion
3. Numerical Pain Rating Scale to assess pain intensity
4. Arabic neck disability index for measuring cervical function

ELIGIBILITY:
Inclusion Criteria:

- 1. Adult subjects aged from 18-35 years old, with FHP using smart phone more than 4 hours per day.

2. Subjects with FHP (craniovertebral angle) [CVA] < 49° 3. Normal body mass index (BMI <25).

Exclusion Criteria:

- 1- Signs of serious pathology (e.g., malignancy, inflammatory disorders, infection).

2- History of cervical spine surgery. 3- History of trauma or fractures in cervical spine. 4- Vascular syndrome such as vertebrobasilar insufficiency.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited from students and employees of Nahda university (smart phone users) from both genders with age ranged between (18-35) years old.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Somatosensory evoked potential of median nerve | at the time of enrollment

SECONDARY OUTCOMES:
change in Craniovertebral angle | At the time of enrollment
Change in cervical range of motion | At the time of enrollment
Change in pain intensity | At the time of enrollment
Assessment of cervical function | At the time of enrollment
  for assessment of cervical function. we will use Neck disability index which is a 10-items questionnaire that measures a patient's self-reported neck pain related disability. Questions include activities of daily living, such as: personal care, lifting, reading, work, driving, sleeping, recreational activities, pain intensity, concentration and headache.

CONTACTS AND LOCATIONS:
Overall Officials: Soheir Shehata Rizkalla, Professor, Study Chair — Department of Basic sciences for physical therapy, Faculty of Physical Therapy , Cairo university, Cairo, Egypt
Locations (1):
- Faculty of Physical Therapy, Nahda University., Bani-Suef, Egypt